CLINICAL TRIAL: NCT02100787
Title: Evaluation of Tear Osmolarity Over Time With Sustained Use of TheraTears Lubricating Drops
Brief Title: Changes in Tear Osmolarity Over Time With Sustained Use of TheraTears
Acronym: BENTLEY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jenkins Eye Care (Other)
Collaborators: Advanced Vision Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVR_PM_102_13
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Dry Eye Syndrome
Keywords: tear osmolarity; keratitis sicca; ocular surface disease; TheraTears
MeSH Terms: conditions — Dry Eye Syndromes; Keratitis sicca

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TheraTears lubricating drops (Experimental): TheraTears lubricating eye drops to be used 1 drop in both eyes four times a day (QID)
  Interventions: Other: TheraTears lubricating drops

INTERVENTIONS:
Other: TheraTears lubricating drops — A over-the-counter lubricating eye drop to be used 1 drop in both eyes 4 times a day (QID) for 8 weeks

SUMMARY:
The objective of the study is to see if there is a change in tear osmolarity over time when moderate to severe dry eye subjects are treated with TheraTears® lubricating drops.

DETAILED DESCRIPTION:
The hypothesis is that the measured tear osmolarity from study participants decrease with sustained use of a over-the-counter artificial tears, TheraTears® lubricating drops, over an eight week period. Participant's dry eye symptoms would also improve with sustained use of TheraTears® lubricating drops.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 21 years of age and has full legal capacity to volunteer;
2. Has read and signed the information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. Is diagnosed with dry eye syndrome (in at least one eye), indicated by current ocular examination, prior history (self-reported history of dry eye is acceptable) and current use of treatments for dry eye;
5. Has a minimum osmolarity reading of 316 mosm/kg at the baseline visit in at least one eye.

Exclusion Criteria:

1. Has taken part in another research study within the last 30 days;
2. Planned contact lens wear during the course of the study;
3. Staff at the investigational site or family member of site staff or family member of currently enrolled participant;
4. Any subject that violates the washout period by using eye drops during the 72hrs washout period;
5. Has any known ocular disease including active ocular infection, inflammation or allergy, especially Salzmann's nodular degeneration, symptomatic conjunctivochalasis, and fixation disparity syndrome;
6. Used Restasis (or similar topical medication) within the last 6 months;
7. Has a systemic condition that in the opinion of the investigator may affect the dry eye status of the subject, especially those newly diagnosed, newly prescribed and/or unstable;
8. Is pregnant, lactating or planning a pregnancy at the time of enrolment (verbal confirmation necessary);
9. Use of medications such as: Systemic Antihistamine (e.g., Allegra®, Benadryl®, Claritin®, Dimetapp®, Unisom®, Zyrtec®, etc.), Isotretinoin (e.g., Accutane®, Roaccutane®, Amnesteem®, Claravis®, Isotroin®, Sotret®) or similar medications;
10. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
11. Has undergone ocular surgery(LASIK, Cataract, etc)within the last year.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-04-10 (Actual); Primary Completion 2016-04-12 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Change in tear osmolarity | Baseline and 8 weeks
Change in the Ocular Surface Disease Index (OSDI) score | Baseline and 8 weeks
  The OSDI is a questionnaire that the subject completes to gauge their dry eye symptoms.

SECONDARY OUTCOMES:
Change in visual acuity | Baseline and 8 weeks
Change in Tear Break Up Time | baseline and 8 weeks
Change in Phenol Red Thread test | baseline and 8 weeks
Change in corneal and conjunctival staining | baseline and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Loretta Ng, OD, Principal Investigator — Jenkins Eye Care
Locations (1):
- Jenkins Eye Care, Honolulu, Hawaii, United States

REFERENCES:
- [Result] Keech A, Senchyna M, Jones L. Impact of time between collection and collection method on human tear fluid osmolarity. Curr Eye Res. 2013 Apr;38(4):428-36. doi: 10.3109/02713683.2013.763987. Epub 2013 Feb 12. PMID 23402632
- [Result] Chia EM, Mitchell P, Rochtchina E, Lee AJ, Maroun R, Wang JJ. Prevalence and associations of dry eye syndrome in an older population: the Blue Mountains Eye Study. Clin Exp Ophthalmol. 2003 Jun;31(3):229-32. doi: 10.1046/j.1442-9071.2003.00634.x. PMID 12786773